CLINICAL TRIAL: NCT04470804
Title: Sirolimus Treatment for Newly Diagnosed Primary Acquired Pure Red Cell Aplasia: a Single Center Prospective Study
Brief Title: Sirolimus Treatment for Newly Diagnosed Primary Acquired PRCA
Acronym: PRCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bing Han (Other)
Responsible Party: Sponsor-Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRCA-2
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pure Red Cell Aplasia, Acquired
Keywords: sirolimus; newly diagnosed pure red cell aplasia; prospective study
MeSH Terms: conditions — Red-Cell Aplasia, Pure | interventions — Sirolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus on newly diagnosed primary acquired PRCA (Experimental): A prospective research of the sirolimus efficiency on newly diagnosed primary acquired PRCA patients. Sirolimus dosage: 2mg QD with plasma concentration 4-15ng/mL. Medication time should last at least 6 months
  Interventions: Drug: Sirolimus
- Cyclosporine A on newly diagnosed primary acquired PRCA (Active Comparator): Cyclosporine A (CsA) efficiency on newly diagnosed primary acquired PRCA patients. CsA dosage: 4mg/kg QD. Medication time should last at least 6 months
  Interventions: Drug: Cyclosporine A

INTERVENTIONS:
Drug: Sirolimus — Sirolimus treats in experimental group
  Other Names: Sirolimus Tablets
  Arms: Sirolimus on newly diagnosed primary acquired PRCA
Drug: Cyclosporine A — Cyclosporine A uses for active comparator group.
  Other Names: Cyclosporine A Tablets
  Arms: Cyclosporine A on newly diagnosed primary acquired PRCA

SUMMARY:
Pure red cell aplasia (PRCA) is a kind of anemia characterized by severe reticulocytopenia and obvious bone marrow erythroblastic cells decreased. Cyclosporine A and /or steroids are the first line therapy but some patients were refractory or intolerance to the treatment. The effects of the second line therapy are also not satisfactory and sometimes not available. The investigators aim to explore the efficacy and side-effect of sirolimus for newly diagnosed primary acquired PRCA.

DETAILED DESCRIPTION:
Pure red cell aplasia (PRCA) is a rare normocytic normochromic anemia with reticulocytopenia, characterized by a reduction of erythroid precursors from the bone marrow, could be divided into congenital and acquired PRCA according to pathogenesis. Congenital PRCA, also known as Diamond-Blackfan syndrome, has been associated with pathogenic variant in GATA1 and TSR2 and gene encode ribosomal proteins. Acquired PRCA can be a primary disease which is usually mediated by immunology, or secondary to other diseases, such as lymphoproliferative diseases, autoimmune diseases, thymoma, infection, or drugs. The first line therapy of acquired PRCA is Cyclosporine A (CsA) and steroids, the second line therapy are anti-CD20, anti-human thymocyte immunoglobulin, immunosuppressive drugs like cyclophosphamide, bone marrow transplantation. Unfortunately, some patients did not response or tolerate the above treatments.

Sirolimus (rapamycin) is an agent produced by the bacterium Streptomyces hygroscopicus, inhibits the mammalian target of rapamycin (mTOR). mTOR is a serine/threonine kinase that regulates cell growth, proliferation, metabolism and survival in eukaryotic cells, and is identified as two interacting complex, mTORC1 and mTORC2. Sirolimus primarily inhibits mTORC1, has been approved for prevent organ transplant rejection, especially in renal transplantation. Sirolimus also promises to treat autoimmune, degenerative and hyperproliferative disorders. Recently, sirolimus has been reported to be effective and well tolerated for many immune-mediated cytopenias, such as autoimmune lymphoproliferative syndrome, immune thrombocytopenia, EVANS syndrome, etc. Some case reports and our previous retrospective study showed that sirolimus was effective for refractory/relapse PRCA with good tolerance. However, due to the rare occurrence of PRCA and good response rate to CsA, there are very few studies of sirolimus on newly diagnosed PRCA so far.

In this study, It is anticipated to evaluate the efficacy and safety of sirolimus versus CsA in patients with newly diagnosed PRCA . The side-effects will be documented and plasma concentration of sirolimus will be monitored. Furthermore, an interim analysis will be performed to assess the treatment efficacy and safety of sirolimus versus CsA in primary PRCA patients when a total of 56 eligible participants finished the designed treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age >18 years old.
2. hemoglobin (Hb) <90 g/L before treatment.
3. no history of immunosuppression therapy prior to sirolimus or CsA treatment.
4. adequate hepatic functions with alanine transaminase (ALT)/aspartate. transaminase (AST) levels within 3 times of the normal upper limit and total bilirubin levels within 2 times of the normal upper limit.
5. documented patient consent.

Exclusion Criteria:

1. diagnosis of secondary aPRCA.
2. history of treatment with immunosuppression therapy before enrollment.
3. history of leukemia, stem cell transplantation, or treatment-related myelodysplastic syndromes (MDS).
4. creatinine/transaminase ≥ 3 normal upper limit.
5. complicated with active or uncontrolled infections or uncontrolled cardiovascular disease.
6. presence of other diseases that may cause anemia.
7. presence of malignancies.
8. pregnant and lactating women.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 6 months
  Hemoglobin level in g/L

SECONDARY OUTCOMES:
Hemoglobin level | 2 years
  Hemoglobin level in g/L

OTHER OUTCOMES:
Overall response | 1 year
  complete response plus partial response
Complete response | 1 year
  Hemoglobin >120 g/L in males or Hemoglobin >110 g/L in females, and lasting for at least 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bride KL, Vincent T, Smith-Whitley K, Lambert MP, Bleesing JJ, Seif AE, Manno CS, Casper J, Grupp SA, Teachey DT. Sirolimus is effective in relapsed/refractory autoimmune cytopenias: results of a prospective multi-institutional trial. Blood. 2016 Jan 7;127(1):17-28. doi: 10.1182/blood-2015-07-657981. Epub 2015 Oct 26. PMID 26504182
- [Result] Li J, Wang Z, Dai L, Cao L, Su J, Zhu M, Yu Z, Bai X, Ruan C. Effects of rapamycin combined with low dose prednisone in patients with chronic immune thrombocytopenia. Clin Dev Immunol. 2013;2013:548085. doi: 10.1155/2013/548085. Epub 2013 Dec 2. PMID 24363761
- [Result] Means RT Jr. Pure red cell aplasia. Blood. 2016 Nov 24;128(21):2504-2509. doi: 10.1182/blood-2016-05-717140. PMID 27881371
- [Result] Teachey DT, Greiner R, Seif A, Attiyeh E, Bleesing J, Choi J, Manno C, Rappaport E, Schwabe D, Sheen C, Sullivan KE, Zhuang H, Wechsler DS, Grupp SA. Treatment with sirolimus results in complete responses in patients with autoimmune lymphoproliferative syndrome. Br J Haematol. 2009 Apr;145(1):101-6. doi: 10.1111/j.1365-2141.2009.07595.x. Epub 2009 Feb 4. PMID 19208097
- [Result] Long Z, Yu F, Du Y, Li H, Chen M, Zhuang J, Han B. Successful treatment of refractory/relapsed acquired pure red cell aplasia with sirolimus. Ann Hematol. 2018 Nov;97(11):2047-2054. doi: 10.1007/s00277-018-3431-5. Epub 2018 Jul 7. PMID 29982851
- [Result] Chen Z, Liu X, Chen M, Yang C, Han B. Successful sirolimus treatment of patients with pure red cell aplasia complicated with renal insufficiency. Ann Hematol. 2020 Apr;99(4):737-741. doi: 10.1007/s00277-020-03946-2. Epub 2020 Feb 6. PMID 32030447
- [Derived] Yang Y, Tang Z, Huang Y, Hu Q, Wang S, Ji J, Du Y, Yang C, Chen M, Hu S, Han B. Sirolimus versus cyclosporine A in patients with primary acquired pure red cell aplasia: a prospective cohort study. Blood Cancer J. 2023 May 10;13(1):74. doi: 10.1038/s41408-023-00845-3. No abstract available. PMID 37160872